CLINICAL TRIAL: NCT00402064
Title: The Influence of Bisphosphonates in the Oral Cavity in Children
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Hadassah Medical Organization, Hadassah Medical Organization
Other Study IDs: st1975-HMO-CTIL
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Oral Cavity; Osteomyelitis; Necrosis of the Jaws
Keywords: bisphosphonates; children; dental; Osteomyelitis; medication
MeSH Terms: conditions — Osteomyelitis

SUMMARY:
The use of bisphosphonates during childhood to ameliorate the skeletal abnormalities associated with osteogenesis imperfecta, idiopathic juvenile osteoporosis, fibrous dysplasia of bone and cerebral palsy. There is paucity of long-term studies among children regarding the safety and efficacy of bisphosphonates.

Osteomyelitis and necrosis of the jaws has been was discovered and reported as a serious adverse event in bisphosphonate-treated adults patients.

To our knowledge, there is no report in the literature about osteomyelitis in children treated with bisphosphonates and the influence of long term treatment with bisphosphonates on children's jaws, the reaction to extractions and on the oral cavity.

Aim of the study: to examine the influence in the oral cavity of bisphosphonate in children

DETAILED DESCRIPTION:
The use of bisphosphonates during childhood to ameliorate the skeletal abnormalities associated with osteogenesis imperfecta, idiopathic juvenile osteoporosis, fibrous dysplasia of bone and cerebral palsy. There is paucity of long-term studies among children regarding the safety and efficacy of bisphosphonates.

Osteomyelitis and necrosis of the jaws has been was discovered and reported as a serious adverse event in bisphosphonate-treated adults patients.

To our knowledge, there is no report in the literature about osteomyelitis in children treated with bisphosphonates and the influence of long term treatment with bisphosphonates on children's jaws, the reaction to extractions and on the oral cavity Aim of the study: to examine the influence in the oral cavity of bisphosphonate in children Materials and methods Population: 50 children treated with bisphosphonate will be included in the study.

The following data will be recorded:

1. age, gender, initial disease, age at diagnosis, additional diseases
2. duration and dosage of the bisphosphonate medication (kind of bisphosphonate, age at the beginning of the drug treatment, duration of treatment, frequency of intake, additional medications)
3. Clinical dental examination was performed for detection of; caries, gingival inflammation and oral hygiene, sequence of dental eruption, teeth extractions, and presence of exposure bone.
4. Unstimulated whole saliva was collected using the spitting method as previously described. Sialochemistry analysis will be performed.
5. Serum analysis findings including: calcium (Ca), phosphorous (P), alkaline phosphatase (AlP) and parathyroid hormone (PTH),vitamin D cross-linked telopeptides (ctx, ntx), bone density. (these examination are performed routinely, in these patients, as part of medical follow up.

ELIGIBILITY:
Inclusion Criteria:

* children treated with bisphosphonate

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children treated with bisphosphonate who attend at the pediatric department of hadassah hospital and or to alyn hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-03; Study Completion 2008-12

CONTACTS AND LOCATIONS:
Overall Officials: diana ram, DMD, Study Director — lecturer, the Hebrew university, Hadassa school of dental medicine
Locations (1):
- Hadassah scool of Dental Medicine, Jerusalem, Israel